CLINICAL TRIAL: NCT02069184
Title: Double Blinded Randomized Placebo Controlled Study in Evaluating the Effectiveness of IV Acetaminophen for Acute Post Operative Pain in C-Section Patients
Brief Title: IV Acetaminophen for Acute Post Operative Pain in C-Section Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Singh Nair, Asst Prof, Anesthesiology, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-07-144
Record Dates: First submitted 2013-12-02; First posted 2014-02-24 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Post-operative Pain
Keywords: opioid usage requirements; pain; IV acetaminophen; opioid usage; c-section
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Acetaminophen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV Acetaminophen (Experimental): IV form, total of 4 doses (each 1000 mg), each every 6th hourly to a maximum dose of 4000 mg in 24 hours.
  Interventions: Drug: IV Acetaminophen
- Saline as placebo (Experimental): IV form, total 4 units, each given every 6th hourly in 24 hours.
  Interventions: Other: Saline as placebo

INTERVENTIONS:
Drug: IV Acetaminophen — 1gm IV. 1st dose at the cord clamping and 3 more doses given every 6th hourly
  Other Names: IV Tylenol
  Arms: IV Acetaminophen
Other: Saline as placebo — 100ml saline IV. 1st dose of 100 ml at cord clamping and 3 more 100ml doses every 6th hourly.
  Arms: Saline as placebo

SUMMARY:
Post-operative pain management after C-section is an important topic as the number of elective c-sections increases each year. Pain is managed either by giving opioids or by using non-opioids. The purpose of this study is to evaluate the effectiveness of IV Acetaminophen in pain relief and its impact in the usage of post-operative opioid requirements and opioid associated complications. The hypothesis is that four doses of IV Acetaminophen in conjunction with intrathecal or epidural morphine given to the patients after c-section will reduce post-operative opioid requirements and opioid associated complications.

DETAILED DESCRIPTION:
Most of the opioids used are centrally acting drugs like morphine or its derivatives. The most common adverse reactions related to systemic administration of opioids are sedation, itching, constipation and less commonly, respiratory depression. One of the other management strategies for the pain control is the use of non-steroidal anti-inflammatory drugs (NSAIDS). Frequent use of NSAIDS is also associated with complications, such as gastric ulcer and platelet dysfunction. When compared to other non-NSAIDS, IV acetaminophen is a relatively safer drug with quicker onset of action. In an earlier conducted study, the onset of action of analgesia for a bolus dose of IV acetaminophen is 3 minutes. IV acetaminophen is FDA approved for management of mild to moderate pain. An adverse reaction associated with the prolonged usage of IV acetaminophen is hepatic injury. The most common adverse events encountered during previous clinical trials were nausea, vomiting, headache and insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Elective full term CS patients
* Age 18 and above
* ASA I-III

Exclusion Criteria:

* Allergic reaction to IV acetaminophen
* Not able to understand and sign the research consent
* Pregnancy induced hypertension or pre-eclampsia patients
* Planned intensive care admission patients
* Patients with severe hepatic impairment or active liver diseases (Two fold increase in any of the liver enzymes)
* Patients with serum creatinine>2mg/dl
* For nursing mothers, any evidence of hepatic dysfunction of the new born

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bernstein, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center- Weiler, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bernstein J, Spitzer Y, Ohaegbulam K, Reddy S, Song J, Romanelli E, Nair S. The analgesic efficacy of IV acetaminophen for acute postoperative pain in C-section patients: a randomized, double-blind, placebo-controlled study. J Matern Fetal Neonatal Med. 2022 Mar;35(5):933-940. doi: 10.1080/14767058.2020.1735337. Epub 2020 Mar 10. PMID 32156175

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Acetaminophen | Saline as Placebo
Started | 33 | 33
Completed | 27 | 31
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen | Saline as Placebo | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31 (6) | 31 (5) | 31 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Opioid Requirements in Cesarean Section (C-section) Patient Population
Time Frame: 24 and 48 hours after Cesarean Section
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | IV Acetaminophen | Saline as Placebo
Number analyzed (Participants) | 33 | 33
mg
  24 hours cumulative | 44 (23) | 48 (28)
  48 hours cumulative | 58 (20) | 57 (22)

2. Secondary Outcome: Visual Analog Score (VAS) Pain Score
Description: Post-operative pain was assessed using VAS pain scores (0-10 scale) with 10 being the worst
Time Frame: every 6 hours for the first 24 hours after the c-section and there after every 8 hours until the patient is discharged or up to 48 hours
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | IV Acetaminophen | Saline as Placebo
Number analyzed (Participants) | 33 | 33
scores on a scale
  0 hr pain after CS | 2.2 (2.9) | 1.4 (2)
  6 hours after CS pain | 3.4 (2.6) | 3.6 (2.5)
  12 hours after CS | 1.2 (1.9) | 2.3 (2.7)
  18 hours after CS | 3.1 (2.7) | 2.9 (3.0)
  24 hours after CS | 4.0 (3.2) | 5.1 (2.1)
  32 hours after CS | 3.1 (2.4) | 2.9 (2.3)
  40 hours after CS | 2.0 (2.2) | 1.2 (1.8)
  48 hours after CS | 3.2 (2.5) | 2.6 (2.1)

3. Secondary Outcome: Percentage of Participants Reporting to be Wide Awake up to 72 Hours After the C-section
Description: Sedation was assessed on a scale of 1-3 (1= wide awake, 2= sleepy but easily aroused, 3= sleepy and difficult to arouse). These assessments were made at the same time points as the pain assessments by the same research assistant. Score 1 is the only good outcome.
Time Frame: Percentage of Participants Reporting to be Wide Awake up to 72 hours after the C-section
Measure: Number; unit: percentage of patients
Arm/Group | IV Acetaminophen | Saline as Placebo
Number analyzed (Participants) | 27 | 31
percentage of patients | 95 | 95

4. Secondary Outcome: "Percentage of Patients With Adverse Events After the Surgery
Description: Subjects were specifically asked about adverse events such as nausea, vomiting, pruritus and breathing difficulties and information regarding their bowel movements. This information was collected on a scale of none, mild, moderate or severe. These are categorical outcomes.
Time Frame: every 6 hours for the first 24 hours after the c-section and there after every 8 hours until the patient is discharged or upto 72 hours. Finally, 1 week after discharge.
Measure: Number; unit: percentage of patients
Arm/Group | IV Acetaminophen | Saline as Placebo
Number analyzed (Participants) | 33 | 33
percentage of patients
  24 hour nausea | 22 | 27
  24 hour vomiting | 21 | 27
  24 hour itching | 57 | 63
  24 hour breathing difficulty | 9 | 6

5. Secondary Outcome: Number of Participants Using Patient-controlled Analgesia (PCA) Attempts
Description: Data were not collected.The use of patient-controlled analgesia (PCA) pumps could have been utilized to standardize rescue medications. This would have allowed the collection of the proportion of subjects that required additional rescue medications. This was another possible endpoint that could have been evaluated.
Time Frame: every 6 hours for the first 24 hours after the c-section and there after every 8 hours until the patient is discharged or upto 72 hours.
Population: None of the participants used PCA pumps so no data could be collected for this outcome measure. PCA was not part of the standard of care at our hospital.
Arm/Group | IV Acetaminophen | Saline as Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants That Were Re-Hospitalized 1 Week After Discharge
Description: No patients were re hospitalized in the first 7 days
Time Frame: From time of discharge to 1 week after discharge
Measure: Number; unit: percentage of patients
Arm/Group | IV Acetaminophen | Saline as Placebo
Number analyzed (Participants) | 33 | 33
percentage of patients | 0 | 0

7. Secondary Outcome: Pain Medication Usage ( NSAIDS)
Description: Compare the percentage of patients using non-opioid pain medication at 24 hours, and 48 hours and had experienced any adverse events.
Time Frame: For the first 24 hours after the c-section until the patient is discharged or up to 48 hours
Measure: Number; unit: percentage of patients
Arm/Group | IV Acetaminophen | Saline as Placebo
Number analyzed (Participants) | 33 | 33
percentage of patients | 27 | 30.3

ADVERSE EVENTS:
Time Frame: 24 hours, 48 hours and up to one week after surgery
Description: Serious and Other (Not Including Serious) Adverse Events
Arm/Group | IV Acetaminophen | Saline as Placebo
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 30/33 | 24/33
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Acetaminophen (N=33) | Saline as Placebo (N=33)
Nausea (Gastrointestinal disorders) | 7 (7) | 7 (7)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Pruritis (Infections and infestations) | 16 (16) | 15 (15)
Breathing Difficulty (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
There may be unknown factors that could have biased the results of the study, pain tolerance is not measured in this study, surgeon variation in performing the surgery and lack of standardized post -operative pain management protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No